CLINICAL TRIAL: NCT00817050
Title: A Preference Evaluation of Nasonex® Nasal Spray (Unscented) vs. Flonase® Nasal Spray (Scented) in Subjects With Symptomatic Allergic Rhinitis (AR) - Single-Dose Cross-over
Brief Title: Single Dose Crossover Study of Patient Preference for Unscented Nasonex® Nasal Spray Versus Scented Flonase® Nasal Spray (Study P04207)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04207
Expanded Access: Available
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasonex Followed by Flonase (Active Comparator)
  Interventions: Drug: Mometasone Furoate Nasal Spray; Drug: fluticasone nasal spray
- Flonase Followed by Nasonex (Active Comparator)
  Interventions: Drug: Mometasone Furoate Nasal Spray; Drug: fluticasone nasal spray

INTERVENTIONS:
Drug: Mometasone Furoate Nasal Spray — One dose (2 sprays in each nostril) of Mometasone Furoate Nasal Spray
  Other Names: Nasonex, SCH 032088
Drug: fluticasone nasal spray — One dose (2 sprays in each nostril) of fluticasone nasal spray
  Other Names: Flonase®

SUMMARY:
This was a one-day single dose trial conducted to compare patient's preference for Nasonex® (mometasone) versus Flonase® nasal spray. Each patient was randomized to take one dose (2 sprays in each nostril) of Nasonex or Flonase. Thirty minutes later, each patient was to take one dose of the opposite medication. Questionnaires were given to each patient after each drug dose to evaluate patient product preference.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been 18-65 years of age, of either sex and any race.
* Subject must have had symptomatic allergic rhinitis with a total nasal symptom (congestion, rhinorrhea, sneezing, itching) severity score of <6 but >2; congestion must have been <2.
* Subject must have been free of any clinically significant disease (other than allergic rhinitis) that would interfere with study evaluations.
* Subject must have understood and been able to adhere to the dosing and visit schedule.

Exclusion Criteria:

* Subject had used any investigational product within 30 days prior to enrollment.
* Subject was in a situation or condition that, in the opinion of the investigator, may have interfered with optimal participation in the study.
* Subject was participating in any other clinical study(ies).
* Subject was using any nasal lavage fluid or spray.
* Subject was using any perfume during the study day.
* Subject was using any oral rinse during the study day.
* Subject had used topical or oral nasal decongestants in the past 1 week.
* Subject had used a nasal corticosteroid in the previous 2 weeks.
* Subject had anosmia or ageusia (absence of the sense of smell or taste).
* Subject had been using medications which are associated with anosmia or ageusia in the 2 weeks prior to testing.
* Subject had a respiratory infection in the 2 weeks prior to testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2005-01-01 (Actual); Study Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
Overall product preference based on subjects' answer to the question "which product do you prefer overall" | On the study day, after dose of each product

SECONDARY OUTCOMES:
Subject rating for likely compliance with daily dosing, | On the study day, after dose of each product
Subject preference for glass or plastic bottle | On the study day, after dose of each product
Subject response to if they would want a prescription for their preferred product and if they would recommend the product | On the study day, after dose of each product
Subject response to whether they preferred inhaled corticosteroid with or without aftertaste, and/or scent/odor, | On the study day, after dose of each product
Subject ratings for individual product attributes | On the study day, after dose of each product